CLINICAL TRIAL: NCT05721690
Title: UED-A Videolaryngoscope vs. Glidescope Titanium for Elective Tracheal Intubation: a Randomized Clinical Trial
Brief Title: UED-A Videolaryngoscope vs. Glidescope Titanium for Elective Tracheal Intubation
Acronym: UED-VLG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Giuseppe Pascarella, Principal Investigator, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAR 72.22
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Intubation; Difficult or Failed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UED-A (Experimental): Tracheal Intubation with UED-A videolaryngoscope
  Interventions: Device: UED-A Videolaryngoscopy
- GLIDESCOPE (Active Comparator): Tracheal Intubation with Glidescope Titanium videolaryngoscope
  Interventions: Device: Glidescope Videolaryngoscopy

INTERVENTIONS:
Device: UED-A Videolaryngoscopy — Tracheal Intubation with UED-A videolaryngoscope
  Arms: UED-A
Device: Glidescope Videolaryngoscopy — Tracheal Intubation with Glidescope Titanium videolaryngoscope
  Arms: GLIDESCOPE

SUMMARY:
The present randomized clinical trial wants to compare the efficacy and safety of UED-A videolaryngoscope to Glidescope Titanium for routinely tracheal intubation in 60 adults, in terms of successful rate, no. attempts and manoeuvre duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidates for general anesthesia in elective general surgery
* Age over 18 years
* American Society of Anesthesiologists (ASA) physical status I-III.

Exclusion Criteria:

* Refusal to sign informed consent
* Paediatric population
* ASA physical status IV
* Emergency tracheal intubation
* Independent Predictors of difficult Videolaryngoscopy (Neck extension < 80°, macroglossia, interincisor distance < 3 cm, anatomical alterations of the neck, cardiac surgery, ear-nose-throat surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-13 (Actual)

PRIMARY OUTCOMES:
Tracheal intubation rate | 30 minutes
  Successful tracheal intubation rate
Number of attempts | 30 minutes
  Number of attempts for a successful tracheal intubation
Total time of intubation | 15 minutes
  Time needed to perform a tracheal intubation from the insertion of the video laryngoscope into the patient mouth
Time to glottis visualization | 15 minutes
  Time needed to visualize the glottis from the insertion of the video laryngoscope into the patient mouth
Cormack-Lehane grade | 15 minutes
  Cormack-Lehane grade observed at videolaryngoscopy Grade 1: Full view of glottis Grade 2: Partial view of glottis Grade 3: Only epiglottis seen, none of glottis seen Grade 4: Neither glottis nor epiglottis seen

SECONDARY OUTCOMES:
Rate of External laryngeal pressure | 15 minutes
  Rate of external laryngeal pressure during laryngoscopy
Rate of of post-laryngoscopy side effects | 24 hours
  Rate of of post-laryngoscopy side effects (bleeding, postoperative sore throat and/or dysphonia)
Rate of Desaturation | 15 minutes
  Rate of Desaturation (spO2 < 93%) during tracheal intubation attempts
Satisfaction Scale | 30 minutes
  Clinicians Satisfaction with the use of the videolaryngoscope, expressed by a 0-10 numeric rating scale (0 = the worst videolaryngoscopy ever performed; 10 = the best videolaryngoscopy ever performed)

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Bio-medico University Hospital Foundation, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agro FE, Doyle DJ, Vennari M. Use of GlideScope(R) in adults: an overview. Minerva Anestesiol. 2015 Mar;81(3):342-51. Epub 2014 May 27. PMID 24861718
- [Background] Law JA, Duggan LV, Asselin M, Baker P, Crosby E, Downey A, Hung OR, Kovacs G, Lemay F, Noppens R, Parotto M, Preston R, Sowers N, Sparrow K, Turkstra TP, Wong DT, Jones PM; Canadian Airway Focus Group. Canadian Airway Focus Group updated consensus-based recommendations for management of the difficult airway: part 2. Planning and implementing safe management of the patient with an anticipated difficult airway. Can J Anaesth. 2021 Sep;68(9):1405-1436. doi: 10.1007/s12630-021-02008-z. Epub 2021 Jun 8. PMID 34105065
- [Background] Aziz MF, Healy D, Kheterpal S, Fu RF, Dillman D, Brambrink AM. Routine clinical practice effectiveness of the Glidescope in difficult airway management: an analysis of 2,004 Glidescope intubations, complications, and failures from two institutions. Anesthesiology. 2011 Jan;114(1):34-41. doi: 10.1097/ALN.0b013e3182023eb7. PMID 21150569
- [Background] Aziz MF, Bayman EO, Van Tienderen MM, Todd MM; StAGE Investigator Group; Brambrink AM. Predictors of difficult videolaryngoscopy with GlideScope(R) or C-MAC(R) with D-blade: secondary analysis from a large comparative videolaryngoscopy trial. Br J Anaesth. 2016 Jul;117(1):118-23. doi: 10.1093/bja/aew128. PMID 27317711
- [Background] Al-Ghamdi AA, El Tahan MR, Khidr AM. Comparison of the Macintosh, GlideScope(R), Airtraq(R), and King Vision laryngoscopes in routine airway management. Minerva Anestesiol. 2016 Dec;82(12):1278-1287. Epub 2016 Apr 22. PMID 27103030
- [Background] Brozek T, Bruthans J, Porizka M, Blaha J, Ulrichova J, Michalek P. A Randomized Comparison of Non-Channeled GlidescopeTM Titanium Versus Channeled KingVisionTM Videolaryngoscope for Orotracheal Intubation in Obese Patients with BMI > 35 kg.m-2. Diagnostics (Basel). 2020 Nov 29;10(12):1024. doi: 10.3390/diagnostics10121024. PMID 33260374
- [Background] Turkstra TP, Turkstra DC, Pavlosky AW, Jones PM. Simultaneous en bloc endotracheal tube insertion with GlideScope(R) Titanium video laryngoscope use: a randomized-controlled trial. Can J Anaesth. 2020 Nov;67(11):1515-1523. doi: 10.1007/s12630-020-01778-2. Epub 2020 Aug 19. PMID 32815101
- [Derived] Migliorelli S, Strumia A, Costa F, Puricelli G, Ruggiero A, Schiavoni L, Mattei A, Carassiti M, Cataldo R, Agro FE, Pascarella G. Hyper-angulated (Glidescope) versus intermediate-angled (UED-A) videolaryngoscopy for routine tracheal intubation in adults: a prospective randomized controlled trial. Sci Rep. 2026 Jan 14;16(1):1986. doi: 10.1038/s41598-025-30932-3. PMID 41535320